CLINICAL TRIAL: NCT03967548
Title: To Evaluate the Local Pharmacokinetic Characteristics of Single Administration of Germinal Peptide Eye Drops in Healthy Volunteers in a Phase I Clinical Study
Brief Title: The Germinal Peptide Eye Drops in Healthy Volunteers in a Clinical Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZK-SFT-201909
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-05

CONDITIONS: Corneal Defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 0.004% single-dose (Experimental): 96 subjects will be treated with Germinal peptide eye drops 0.004% single dose (16 were pre-tested and 64 were formally tested).
  Interventions: Drug: Germinal peptide eye drops

INTERVENTIONS:
Drug: Germinal peptide eye drops — Germinal peptide eye drops of 0.004%
  Other Names: shengfatai-eye drops

SUMMARY:
The subjects of this study were healthy subjects, who were given medicine in a single dose group: 0.004%.

DETAILED DESCRIPTION:
Tear collection was conducted on the single dose D1 (that is, the day of administration). Collection points: 10 min, 30 min, 1 h, 2 h, 4 h, 6 h, 8 h, and 12 h after administration.Each time 5-50 mg (generally 20 mg), a total of 160-1600 mg of tears will be collected (during the screening period, all subjects will retain the tear samples collected by the Schirmer filter paper, among which, qualified tear samples will be used for blank samples or methodological investigation.After administration, only 1 tear collection site will be collected for each subject.

ELIGIBILITY:
Inclusion Criteria:

1. healthy volunteers aged between 18 and 45, both male and female in each group;
2. body mass index between 19 and 26 kg/m2 (including critical value), male weight 50 kg, female weight 45 kg;
3. target eye Schirmer Ⅰ test (Schirmer filter paper bending, clip next eyelid medial 1/3 conjunctival sac within 5 min) tear wet filter paper length or greater 10 mm;
4. subjects will participate in the study voluntarily and sign the informed consent.

Exclusion Criteria:

1. binocular corrected vision < 1.0, abnormal intraocular pressure, slit lamp and fundus examination with clinical significance;
2. those with abnormal physical examination, vital signs, electrocardiogram and laboratory examination before the test with clinical significance;
3. patients with eye diseases, including history of inner eye surgery or laser surgery;
4. a medical history of central nervous system, spirit, cardiovascular system, kidney, liver, respiratory system, metabolism system and skeletal muscle system, which may endanger the safety of subjects or affect the results of the study;
5. positive test results of hepatitis b virus surface antigen (HBsAg), hepatitis c virus antibody (hcv-ab), treponema pallidum specific antibody (tp-ab) or human immunodeficiency virus antibody (hiv-p24 /Ab);
6. have a significant history of clinical allergy, especially drug allergy, especially allergic to any component of germinal peptide eye drops;
7. smoking more than 5 cigarettes per day on average;
8. those who are suspected or have alcohol dependence, and their alcohol intake is more than 2 units per day on average for 3 months (1 unit =10 mL ethanol, that is, 1 unit =200 mL beer with 5% alcohol or 25 mL spirit with 40% alcohol or 83 mL wine with 12% alcohol) or who have tested positive for alcohol;
9. history of drug abuse, or positive urine test of ketamine, morphine, methamphetamine, dimethylene dioxyamphetamine, tetrahydrocannabinic acid;
10. have taken any medicine within 2 weeks before screening;
11. participated in clinical trials within the first 3 months of screening;
12. blood donation or blood loss 400 mL within 3 months before screening;
13. have used ophthalmic drugs or eyelash growth solution in the first 2 weeks;
14. select the subjects who have worn contact lenses or contact lenses in the first 2 weeks;
15. pregnant or lactating women and those planning to become pregnant (including male subjects);No effective contraceptive measures were taken within 1 month prior to the inclusion of subjects, or subjects (including male subjects) were unwilling to take effective contraceptive measures within the next 6 months;
16. the researchers considered the participants unsuitable.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-05-16 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Area under curve （0-t） | Within 12hours after administration
  AUC（0-t）
Area under curve（0-∞） | Within 12hours after administration
  AUC（0-∞）
Peak concentration | Within 12hours after administration
  Cmax
Peak time | Within 12hours after administration
  Tmax
Half life | Within 12hours after administration
  t1/2
Apparent volume of distribution | Within 12hours after administration
  Vd
Elimination rate constant | Within 12hours after administration
  Kel
Mean residence time | Within 12hours after administration
  MRT
Clearance | Within 12hours after administration
  CL or CL/F

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zhao, PHD, Study Director — Beijing Tongren Hospital
Locations (1):
- Xiuli Zhao, Beijing, China